CLINICAL TRIAL: NCT01673620
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety of Combination Montelukast/Loratadine (MK-0476A) in Mexican Patients With Allergic Rhinitis
Brief Title: A Study to Evaluate the Safety of Combination Montelukast/Loratadine in Mexican Participants With Allergic Rhinitis (MK-0476A-484)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476A-484
Record Dates: First submitted 2012-08-03; First posted 2012-08-28 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2024-09-04 (Actual); Status verified 2022-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — montelukast; Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast 10 mg/loratadine 10 mg (Experimental): Montelukast 10 mg/loratadine 10 mg combination tablet administered orally once daily for 2 weeks
  Interventions: Drug: Montelukast 10 mg/loratadine 10 mg
- Placebo (Placebo Comparator): Matching placebo tablet administered orally once daily for 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast 10 mg/loratadine 10 mg — Montelukast 10 mg/loratadine 10 mg tablet administered once daily
  Other Names: MK-0476A
  Arms: Montelukast 10 mg/loratadine 10 mg
Drug: Placebo — Matching placebo tablet administered once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of montelukast 10 mg/loratadine 10 mg versus placebo in Mexican participants with allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant or breastfeeding and does not plan to become pregnant during the study and the 14-day follow-up period
* Female participants of reproductive potential agree to remain abstinent or use one acceptable method of birth control at least 14 days prior to signing the informed consent until 14 days following the last visit
* History for at least 2 years of seasonal allergic rhinitis symptoms that are known to flare during the local allergy season or a clinical history of at least 2 years of perennial allergic rhinitis symptoms that persist year round
* For participants with seasonal allergic rhinitis: a positive skin-prick test (wheal >= 3 mm greater than saline control) to one of the allergens active during the local allergy season or a positive radioallergosorbent test (RAST [defined as a score >= Class III])
* For participants with perennial allergic rhinitis: a positive skin test (wheal >=3 mm greater than saline control) to one of the relevant perennial allergens or a positive RAST (defined as a score >= Class III)
* Nonsmoker and has been a nonsmoker for at least 1 year prior to study Visit 1 with a smoking history of no more than 10 pack-years (1 pack [20 cigarettes] per day for 10 years)
* Must be in good and stable physical health and mental health

Exclusion Criteria:

* Hospitalization or hospitalization within 4 weeks of the first scheduled study visit
* Pregnancy or within <= 8 weeks postpartum or is breast feeding
* Any major surgical procedure within 4 weeks of the first scheduled study vist
* Current or recent past abuser of alcohol or illicit drugs
* Prior participation in a clinical trial of montelukast or loratadine within the 4 weeks prior to the first scheduled study visit
* Requires treatment other than inhaled short-acting β-agonist for asthma

  (e.g., inhaled or oral corticosteroid, theophylline, nedocromil, cromolyn, oral or long-acting inhaled β-agonist, leukotriene receptor antagonist, leukotriene synthesis inhibitor) and/or uses more than 8 puffs per day of inhaled short-acting β-agonist
* Presence of an upper respiratory tract infection (URI), sinusitis, infectious rhinitis (with symptoms such as sore throat, fever, thick purulent rhinorrhea), ocular infection, or history of any of these within 4 weeks prior to the first scheduled study visit or any time between study Visits 1 and 2
* Other than asthma, any active, acute, or chronic pulmonary disorder which is documented by history or physical examination
* Rhinitis medicamentosa, or non-allergic rhinitis
* Recent history (within 3 months prior to the first scheduled study visit) of a clinically significant psychiatric disorder
* History of an anaphylactic reaction to or is otherwise hypersensitive to

montelukast, loratadine, or one of their components

* History or current evidence of any general medical condition, concomitant therapy, lab abnormality or other circumstance that might confound the results of the study or interfere with the patient's participation for the full duration of the study
* History of illness that would require treatment with an excluded medication, could be immediately life threatening (ventricular arrhythmia, diabetes mellitus that is not well controlled), would pose restriction on participation or successful completion of the study, or would pose additional risk to the patient by administering the study drug
* History of malignancy ≤5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-07-04 (Actual); Primary Completion 2012-10-10 (Actual); Study Completion 2012-10-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Montelukast 10 mg/Loratadine 10 mg: Participants receive montelukast 10 mg/loratadine 10 mg combination tablets once daily for 2 weeks
- Placebo: Participants receive matching placebo tablets once daily for 2 weeks
Period: Overall Study
Arm/Group | Montelukast 10 mg/Loratadine 10 mg | Placebo
Started | 47 | 22
Completed | 46 | 22
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast 10 mg/Loratadine 10 mg | Placebo | Total
Number analyzed (Participants) | 47 | 22 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (12.5) | 31.9 (9.3) | 30.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 14 | 44
  Male | 17 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing at Least One Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study treatment, whether or not considered related to the use of the study treatment.
Time Frame: Up to 4 weeks
Population: The All-Patients-as-Treated (APaT) population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Montelukast 10 mg/Loratadine 10 mg | Placebo
Number analyzed (Participants) | 47 | 22
participants | 6 | 2

2. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to AEs
Description: as for outcome 1
Time Frame: Up to 2 weeks
Population: The APaT population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Montelukast 10 mg/Loratadine 10 mg | Placebo
Number analyzed (Participants) | 47 | 22
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Description: The APaT population consisted of all randomized participants who received at least one dose of study drug.
Arm/Group | Montelukast 10 mg/Loratadine 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/22
Other Adverse Events (participants affected / at risk) | 3/47 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast 10 mg/Loratadine 10 mg (N=47) | Placebo (N=22)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.